CLINICAL TRIAL: NCT05877638
Title: Randomized Controlled Trial Assessing a Novel Glycopolymer Compound in the Treatment of Superficial Partial-Thickness Burns
Brief Title: SWC for Treatment of Superficial Partial-Thickness Burns
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Synedgen, Inc. (Industry)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWC
Record Dates: First submitted 2023-03-27; First posted 2023-05-26 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-05

CONDITIONS: Burn Wounds
MeSH Terms: conditions — Burns | interventions — Silver Sulfadiazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SynePure with Catasyn (Experimental): SynePure Wound Cleanser and Catasyn Advanced Technology Hydrogel
  Interventions: Device: SynePure Wound Cleanser and Catasyn Advanced Technology Hydrogel
- Silvadene (Active Comparator): Routine care wound rinse and Silvadene cream
  Interventions: Drug: SILVADENE Cream 1% (silver sulfadiazine)

INTERVENTIONS:
Device: SynePure Wound Cleanser and Catasyn Advanced Technology Hydrogel — (FDA) 510(k) cleared wound care medical devices formulated with a novel biocompatible chitosan derivative, poly (acetyl, arginyl) glucosamine. SynePure is optimized for the cleansing and debridement of wounds and thermal injuries, and Catasyn serves as a protective gel dressing.
  Arms: SynePure with Catasyn
Drug: SILVADENE Cream 1% (silver sulfadiazine) — SILVADENE Cream 1% (silver sulfadiazine) is a topical antimicrobial drug indicated as an adjunct for the prevention and treatment of wound sepsis in patients with second- and third-degree burns.
  Arms: Silvadene

SUMMARY:
The purpose of this study is to test the safety and effectiveness of SynePure™ Wound Cleanser when used in combination with Catasyn™ Advanced Technology Hydrogel for the treatment of superficial partial-thickness burn wounds.

DETAILED DESCRIPTION:
Current management options for burn wounds contain silver (nanoparticulate or ionic), hypochlorite, hydrogen peroxide, sulfa agents, chlorhexidine, iodine or other dilute antiseptics meant to provide some measure of antimicrobial protection. However, all of these materials have some proven limitations in facilitating wound healing and also have notable local and systemic adverse effects. None of the current clinical treatments enhance healing and/or reduce scar formation. The purpose of this study is to test the safety and effectiveness of SynePure™ Wound Cleanser when used in combination with Catasyn™ Advanced Technology Hydrogel for the treatment of superficial partial-thickness burn wounds.

This study is a prospective, parallel group, randomized controlled trial comparing SynePure Wound Cleanser and Catasyn Advanced Technology Hydrogel (intervention group) to routine care, Silvadene (control group). Both groups will receive the same care other than the treating agent. Subjects will be recruited from the Burn Center/Clinic adult patient pool who have sustained superficial partial-thickness burn wounds that comprise ≤15% of total body surface area (TBSA).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have sustained superficial, partial thickness burn wounds no less than 5% and up to 15% of total body surface area (TBSA; 5-15%). Contiguous superficial and deep partial-thickness burns are eligible for inclusion.
* Patients otherwise in good general physical and mental health, as per the investigator's clinical judgment.

Exclusion Criteria:

* Inability to provide informed consent
* Deep partial-thickness burns except as noted in the inclusion criteria and full-thickness burns
* Radiation, chemical or electrical burn injury
* Patients with burns primarily located to the face, genitals, or span across joints
* Patients whose burn injury was ≥ 8 days prior to entry into the Burn Center/ Clinic.
* Patients with uncontrolled cerebrovascular disease, cardiovascular disease, concurrent endocrine, hepatic or renal disease, or other severe conditions for whom, in the investigators' discretion would render study participation unsafe
* Patients with documented or self-reported shellfish allergies
* Current pregnancy
* Patients with concurrent burn related injuries or inhalation injury that would put the patient at increased risk, per physician discretion
* Any condition to which in the investigator's discretion would render study enrollment a safety concern for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Percentage of healing wound progress across study window | Up to 21days
  Healing is defined as 90% re-epithelialization (skin and mucous membrane replacement) of the wounded area

SECONDARY OUTCOMES:
Number of new infection rates | Up to 21days
  Characterized by local new inflammation, heat, purulence as well as new or increased pain, redness and swelling

OTHER OUTCOMES:
Number of complications other than infection | Up to 21days
  Complications such as gangrene, necrosis, periwound dermatitis and/or edema, hematoma, or any other complication determined to be related to the wound and/or treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shenda Baker, PhD, Principal Investigator — Synedgen, Inc.
Locations (1):
- Louisiana State University Health Science Center at New Orleans, New Orleans, Louisiana, United States